CLINICAL TRIAL: NCT01100359
Title: Phase II Multicenter Trial of the Austrian AGO With the Combination of Liposomal Doxorubicin (Myocet®) and Carboplatin in Primary Advanced or Metastatic and Recurrent Endometrial Cancer
Brief Title: Liposome-Encapsulated Doxorubicin Citrate and Carboplatin in Treating Patients With Advanced or Metastatic Recurrent Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: MUI-AGO-15; CDR0000669712 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2007-004060-40; EU-21027
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2011-02

CONDITIONS: Endometrial Cancer
Keywords: endometrial clear cell carcinoma; recurrent endometrial carcinoma; stage IIIA endometrial carcinoma; stage IIIB endometrial carcinoma; stage IIIC endometrial carcinoma; stage IVA endometrial carcinoma; stage IVB endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin

INTERVENTIONS:
Drug: carboplatin
Drug: liposome-encapsulated doxorubicin citrate
Other: laboratory biomarker analysis
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposome-encapsulated doxorubicin citrate and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well liposome-encapsulated doxorubicin citrate given together with carboplatin works in treating patients with advanced or metastatic recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess activity of the combination of liposome-encapsulated doxorubicin citrate and carboplatin in patients with primary advanced or metastatic recurrent carcinoma of the endometrium.

Secondary

* To assess the toxicity and feasibility of this regimen in these patients.
* To determine the progression-free survival and overall survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive liposome-encapsulated doxorubicin citrate IV over 1 hour followed by carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 6-9 courses in the absence of disease progression or unacceptable toxicity.

Tissue array and immunohistochemistry analysis are conducted on paraffin-embedded tumor blocks of the primarily operated tissue of all patients for different markers (e.g., progesterone-/estrogen receptor, HER2-receptor, soluble L1-molecule, Topo 2a) to examine tumor characteristics.

Quality of life is assessed at baseline, during study treatment, at completion of study treatment, and then at 1 year after completion of study treatment.

After completion of study therapy, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of endometrial carcinoma, including any of the following cellular types:

  * Mixed Mullerian carcinoma
  * Serous carcinoma
  * Clear cell carcinoma
* Primary advanced (FIGO stage III or stage IV) or metastatic recurrent disease
* Disease not curable by surgery
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm with x-ray, physical exam, or non-spiral CT scan OR ≥ 10 mm with spiral CT scan or MRI
* No known cerebral metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 100,000/mm^3
* ANC ≥ 1,500/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.25 times upper limit of normal (ULN)
* Bilirubin ≤ 1.25 times ULN
* AST/ALT < 3 times ULN
* Glomerular filtration rate ≥ 50 mL/min
* LVEF ≥ 50% by ECHO
* Fertile patients must use effective contraception
* No myocardial infarction within the past 6 months
* No NYHA class II-IV congestive heart failure
* No third degree or complete heart block unless a pacemaker is in place
* No other malignancy within the past 5 years
* No concomitant medical illness (e.g., uncontrolled infection, uncontrolled angina, or other relevant illness) that makes the prescribed treatments within this study unfeasible
* No known hypersensitivity to study drugs
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for disease recurrence
* At least 12 months since prior adjuvant therapy containing anthracyclines with cumulative doses not exceeding the following:

  * Epirubicin 600 mg/m²
  * Doxorubicin 300 mg/m²
* At least 6 months since prior adjuvant therapy containing platinum
* At least 4 weeks since completion of radiotherapy involving the whole pelvis
* No concurrent radiotherapy or planned radiotherapy after study
* No concurrent endocrine, immunological, or other anticancer therapy
* No concurrent participation in another investigational drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Duration of progression-free survival
Overall survival
Safety
Feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Christian Marth, MD, PhD, Study Chair — Medical University Innsbruck
Locations (1):
- Innsbruck Universitaetsklinik, Innsbruck, Austria